CLINICAL TRIAL: NCT06705075
Title: Evaluation of Uterine Fibroids by Contrast Enhanced Ultrasound (CEUS) and Subharmonic- Aided Pressure Estimation (SHAPE) Pre and Post-Uterine Artery Embolization (UAE)
Brief Title: Evaluation of Uterine Fibroids by CEUS and SHAPE Pre and Post UAE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Priscilla Machado, Research Assistant Professor, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: iRISID-2024-0851
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-11

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Uterine fibroids (Experimental)
  Interventions: Drug: Perfluten

INTERVENTIONS:
Drug: Perfluten — Use of UCA Definity to evaluate uterine fibroids by contrast-enhanced ultrasound (CEUS) and subharmonic-aided pressure estimation (SHAPE) pre and post-uterine artery embolization (UAE).

SUMMARY:
This study goals are to determine the patterns of uterine fibroid vascularity pre and post UAE using CEUS resulting in an alternative to gadolinium-enhanced MRI that is less expensive, has less contra-indications and side effects, is real time, and noninvasive helping physicians to evaluate the result of UAE procedures. Also, this study will evaluate uterine fibroid pressures using SHAPE, comparing the results with normal myometrium tissue in order to determine its characteristics and tissue differences, which we believe will lead to the development of a new biomarker for the diagnosis and treatment of uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Be a female diagnosed with endometrial cancer and scheduled for UAE.
* Be over the age of 18 years.
* If the subject is of child-bearing potential, must have a negative pregnancy test.
* Be conscious and able to comply with study procedures.
* Have read and signed the IRB approved consent form for participating in the study.

Exclusion Criteria:

* Females who are pregnant or nursing.
* Patients who have received an investigational drug in the 30 days before study drug administration, or will receive one within 72 hours afterwards.
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable. For example:
* Patients on life support or in a critical care unit.
* Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia.
* Patients with recent cerebral hemorrhage.
* Patients who have undergone surgery within 24 hours prior to the study sonographic examination.
* Patients with congenital heart defects.
* Patient with a known allergy to Definity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Uterine Fibroids by Contrast Enhanced Ultrasound (CEUS) and Subharmonic- Aided Pressure Estimation (SHAPE) Pre and Post-Uterine Artery Embolization (UAE). | 2 years
  This is an open-label, non-randomized, single center, clinical study that will be conducted at TJU. This trial of CEUS and SHAPE imaging examinations will evaluate the microvascularity of uterine fibroids in order to determine vascularity characteristics before,2 weeks, as well as 3 months after UAE to assess the success of the UAE procedure in short term follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided